CLINICAL TRIAL: NCT02805140
Title: The Moms Online Video Exercise Study
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Maya Mascarenhas, MPH, Doctoral Student, Epidemiology & Biostatistics, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-15344
Record Dates: First submitted 2016-03-28; First posted 2016-06-17 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Sedentary Lifestyle
Keywords: mother; social support; mobile app; videoconference; sedentary; physical activity
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual exercise and mobile apps (Experimental): Participants randomized to the intervention arm will join a virtual group convenient for them. They will plan and participate in 8 weeks (every week day) of virtual exercise sessions. Sessions will all be under 30 minutes and include a brief check in amongst participants. The investigators will provide links to information on physical activity and links to online resources for being active.
  Interventions: Behavioral: Virtual exercise; Behavioral: Mobile apps; Behavioral: Exercise resources and information
- Exercise resources and information (Active Comparator): The investigators will provide links to information on physical activity and links to online resources for being active. Women will be invited to join the exercise groups at the end of the 8 weeks.
  Interventions: Behavioral: Exercise resources and information

INTERVENTIONS:
Behavioral: Virtual exercise — Using videoconferencing, mothers assigned to intervention arm will participate in daily (weekdays) virtual exercise sessions for 6 weeks with other mothers.
  Arms: Virtual exercise and mobile apps
Behavioral: Mobile apps — During virtual exercise sessions, mothers assigned to intervention arm will follow exercise routines using mobile exercise apps that are recommended by study staff.
  Arms: Virtual exercise and mobile apps
Behavioral: Exercise resources and information — For all mothers, the investigators will provide standard information on the benefits of exercise and link to existing public health resources on how to start and stay active.

SUMMARY:
The purpose of this study is to test feasibility and acceptability of an online platform that uses mobile apps and videoconferencing tools to increase activity levels in mothers with young children.

DETAILED DESCRIPTION:
The investigators are testing the feasibility and acceptability of a digital health platform using a randomized parallel wait-list control design for mothers with young children. The platform incorporates home based supportive group exercise sessions using video conferencing tools, shared online activity tracking and exercise mobile apps for individualized exercise routines will help mothers increase their physical activity levels and be successful at maintaining this increase.

The intervention arm consists of two main parts: home based video conferencing virtual exercise sessions and mobile exercise apps, which women use to tailor exercise routines to their own skill level and preferences. Both arms will receive an activity monitor that they collect continuous activity data throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Mother to at least one child that is less than 18 years old
* Owns a smart phone (iPhone or Android) and can download mobile applications
* Sufficient data to use mobile applications on a mobile device
* Owns a mobile device with a web camera

Exclusion Criteria:

* Inability to provide informed consent
* Inability to speak or understand English
* Any medical restrictions where vigorous activity is not recommended
* Any history of heart conditions including cardiovascular disease or coronary artery disease
* Any history of heart conditions including cardiovascular disease or coronary artery disease
* Meets federal guidelines for exercise for either aerobic (150 minutes of moderate activity per week, 75 minutes of vigorous activity per week, or some combination)
* Pregnant or planning to get pregnant during study duration

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment | End of 8 week recruitment period
  Recruiting 75% of goal of 38 participants
Acceptability of study procedures | End of 8 week intervention period
  We will consider at least 75% of participants being "satisfied" or "very satisfied" (using a Likert scale) in the overall study evaluation to indicate acceptability of the study materials.
Change in minutes per week of moderate-to-vigorous physical activity | 0 weeks, 8 weeks
  Active minutes (past 7 days) using self report through Active Australia Survey

SECONDARY OUTCOMES:
Change in exercise self efficacy | 0 weeks, 8 weeks
  Using Sallis Short Form 3 item self efficacy scale, the investigators will measure changes in exercise self efficacy
Change in exercise enjoyment | 0 weeks, 8 weeks
  Using Sallis Short Form 3 item exercise enjoyment scale, the investigators will measure changes in exercise enjoyment
Change in exercise social support | 0 weeks, 8 weeks
  Using Sallis Short Form 3 item exercise social support scale, the investigators will measure changes in exercise social support
Change in global health | 0 weeks, 8 weeks
  Using NIH Patient Reported Outcome Measurement System (PROMIS) Global Health 7 item measure, the investigators will measure overall changes in global health
Change in fatigue | 0 weeks, 8 weeks
  Using NIH Patient Reported Outcome Measurement System (PROMIS) Global Health 4 item measure, the investigators will measure overall changes in fatigue
Change in weight | 0 weeks, 8 weeks
  Difference in pounds gained or lost in lbs measured by self report via survey

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mascarenhas MN, Chan JM, Vittinghoff E, Van Blarigan EL, Hecht F. Increasing Physical Activity in Mothers Using Video Exercise Groups and Exercise Mobile Apps: Randomized Controlled Trial. J Med Internet Res. 2018 May 18;20(5):e179. doi: 10.2196/jmir.9310. PMID 29776899